CLINICAL TRIAL: NCT01713296
Title: A Phase II Trial of Pazopanib, in Relapsed and Refractory Small Cell Lung Cancer (SCLC)
Brief Title: Pazopanib in Relapsed and Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/11.01
Record Dates: First submitted 2012-09-27; First posted 2012-10-24 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: SCLC
Keywords: SCLC; 2nd Line; Relapsed or Refractory
MeSH Terms: conditions — Recurrence | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental)
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Pazopanib: 800mg once a day for up to 2 years from date of first dose

SUMMARY:
Investigators propose to study the single agent activity of pazopanib in a Phase II trial of patients with relapsed or refractory small cell lung cancer. Because these patients have very limited treatment options, use of an investigational agent in this patient population is supported by current National Comprehensive Cancer Network guidelines. Using correlative biologic studies to evaluate the anti angiogenic activity of pazopanib in the absence of concomitant chemotherapy will allow us to delineate the responses due to this drug and the effect on angiogenesis.

Pazopanib dose has been determined to 800 mg once daily per the initial recommended dose approved by FDA and EMA, as monotherapy in advanced Renal Cell Carcinoma

DETAILED DESCRIPTION:
Small cell lung cancer is a tumor that initially responds to chemotherapy and radiotherapy, however, it is associated with very poor prognosis since the initial response is nearly always followed by relapse and metastasis. The response to subsequent therapy is very limited as is the duration of response in these patients. Patients with SCLC have high rates of metastases at presentation suggesting that angiogenesis is particularly important in this cancer, furthermore studies have shown that microvessel density and VEGF expression in SCLC tumor samples correlate with development of metastases and poor prognosis. Furthermore VEGF expression was the only factor that retained a significant inverse correlation with survival when assessed in a multivariate analysis.

Pazopanib is a potent, small molecule competitive inhibitor of the tyrosine kinase activity of (VEGFR 1), VEGFR 2, VEGFR 3, platelet derived growth factor (PDGF), and c kit, capable of inhibiting downstream signalling from these receptors. The IC50 of pazopanib against VEGFR 2 is 10nm, and the IC50 against VEGFR 1 is <50nm. Currently a number of studies is underway for the evaluation of pazopanib in the treatment NSCLC. Administering pazopanib to patients with relapsed SCLC offers an attractive choice in patients with very limited therapeutic choices. The high rate of metastasis highlights the need for alternative treatments that act directly on the growth and invasion of tumors and subsequent development of metastases, rather than solely on cell proliferation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up Procedures conducted as part of the patient's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Age ≥ 18 years
* Diagnosis of SCLC based on either histology or cytology (by FNA) with radiologically confirmed progressive disease after first-line chemotherapy.
* Presence of brain metastases is permitted if patient has completed treatment with surgery and/or radiation more than four weeks prior to date of first dose of study drug. Patients who have developed brain metastases following prophylactic cranial irradiation will not be eligible for participation
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Measurable disease criteria according to RECIST 1.1
* Only one prior chemotherapy regimen
* Biologic material (blood samples, archived tissue) will be collected from consenting patients for biomarker analysis before and/or during treatment with investigational product
* Adequate organ system function
* Localised irradiation for SCLC is permitted as long as it was a minimum of 4 weeks before entering the study; however, single-dose palliative radiation of bone metastases for pain control may be allowed during the 4-week screening period
* A female is eligible to enter and participate in this study if she is of:

Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had: A hysterectomy, A bilateral oophorectomy (ovariectomy), A bilateral tubal ligation, Is post-menopausal

* Patients not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L)
* Patients using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow: Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product. Oral contraceptive, either combined or progestogen alone. Injectable progestogen.Implants of levonorgestre. Estrogenic vaginal ring. Percutaneous contraceptive patches. Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year. Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository) Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug

Exclusion Criteria:

* Prior malignancy
* Prior use of an investigational or licensed drug that targets VEGF or VEGF receptors
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:
* Active peptic ulcer disease
* Known intraluminal metastatic lesion/s with risk of bleeding
* Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: Malabsorption syndrome, Major resection of the stomach or small bowel
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting, Myocardial infarction, Unstable angina, Coronary artery bypass graft surgery, Symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg]
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary haemorrhage, for example: Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed, Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed, Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, tumour touching but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions)
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
* Treatment with any of the following anti-cancer therapies: radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib or chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Rate | 2 Years
  Patients will be assessed every 8 weeks, from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 168 weeks

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Patients overall survival will be calculated from the date of the first chemotherapy cycle until the date of death from any cause
Toxicity profile | Every 4 weeks
  Patients will be evaluated on Day 1 of each cycle (cycle repeated every 4 weeks)up to two years from the date of first dose administration

CONTACTS AND LOCATIONS:
Locations (8):
- Greece (8):
  - "Agioi Anargyroi" Anticancer Hospital of Athens, Athens
  - "IASO" General Hospital of Athens, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Papageorgiou" Hospital of Thessaloniki, Thessaloniki
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki